CLINICAL TRIAL: NCT05368155
Title: Chronic Pelvic Pain and Education Skills Training for Women Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Derrecka Boykin, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-51197
Record Dates: First submitted 2022-05-03; First posted 2022-05-10 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Pain; Depression, Anxiety
Keywords: Acceptance and Commitment Therapy; Women Veterans; Primary Care
MeSH Terms: conditions — Pelvic Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT and Education Group (Experimental): The Acceptance and Commitment Training (ACT) and education group will receive the Brief ACT for Pelvic Pain treatment, which will include three weekly, 90-minute group sessions.
  Interventions: Behavioral: Brief ACT for Pelvic Pain
- Enhanced Treatment As Usual (No Intervention): The Enhanced treatment as usual (TAU) condition will receive a letter with treatment resources and encouraged to consult with their VHA primary care clinicians for additional education and treatment options.

INTERVENTIONS:
Behavioral: Brief ACT for Pelvic Pain — The Brief ACT for Pelvic Pain treatment will include three weekly, 90-minute group sessions that teach Veterans new ways to respond to difficult thoughts and emotions related to pain (Acceptance and Mindfulness Training) and encourage behavioral (re)engagement in meaningful life activities (Behavioral Change Training). The overall goal is to cultivate psychological flexibility by helping Veterans learn to respond to life events in ways which do not exacerbate difficulties or restrict engagement in meaningful activities. Workshop content is integrated with education on pelvic pain (its diagnostic criteria, etiology, and associated health outcomes) to increase alignment of the treatment with patient needs.
  Arms: ACT and Education Group

SUMMARY:
Chronic pelvic pain (CPP) is a debilitating condition that disproportionately affects women Veterans (25% vs. 16% of civilian women). Predisposing factors include higher rates of strenuous physical activity during military service, duty-related injuries, psychiatric distress, and sexual trauma. CPP is associated with a high burden of illness, disability, and economic costs (estimated at $5.8 billion in annual health care expenditures).

Multimodal, interdisciplinary approaches are emphasized in the treatment of CPP. Psychological interventions are essential for optimizing pain self-management for CPP. Psychosocial factors are known to affect pain intensity and recovery. Women Veterans report higher rates of depression and anxiety with CPP, that leads to greater disability and poorer quality of life. Cognitive and behavioral therapies, such as Acceptance and Commitment Therapy (ACT), are effective options for pain self-management. Barriers to effective pain treatment are high attrition and non-adherence. Additionally, women Veterans prefer treatments that address their gender-specific needs. Gender-specific services remain limited in the Veterans Health Administration (VHA).

In line with VHA's priorities to expand women's health care, this study implements ACT in a brief intervention format to address a highly prevalent reproductive health issue among women Veterans. ACT is transdiagnostic and thus provides a unified approach to the treatment of co-occurring disorders, such as chronic pain, depression, and anxiety. Brief workshop formats increase treatment completion and patient engagement. This study seeks to adapt an existing 1-day ACT workshop for use in VHA integrated primary care (PCMHI) and specialty medical settings with women veterans experiencing CPP. Primary outcomes are feasibility and acceptability of the adapted intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being a Veteran
* Being female
* Having a diagnosis of chronic pelvic pain
* Endorsing severe pain (score ≤ 7 on Brief Pain Inventory [BPI]) or moderate to severe pain plus clinically significant psychological distress (score ≤ 3 on BPI and score ≤ 10 on Patient Health Questionnaire-9 [PHQ-9] or Generalized Anxiety Disorder-7 [GAD-7])

Exclusion Criteria:

* Cognitive impairment
* An uncontrolled bipolar or psychotic diagnosis
* Active suicidal ideation
* Receiving concurrent psychotherapy or who have received ACT within the past year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only participants who identify as "female" can take part in this study. The intervention is specifically designed for women veterans who experience chronic pelvic pain.
Enrollment: 13 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | Up to 1 year
  Recruitment rates (number enrolled/number who complete treatment)
Acceptability of intervention | 2-month follow-up
  Open-ended question about how satisfactory veterans find the intervention (including likes, dislikes, and recommendations for improving the intervention)

SECONDARY OUTCOMES:
Mean change score in Patient Health Questionnaire (PHQ-9) | Change at 2-month follow-up from baseline
  The 9-item PHQ-9 measures severity of depressive symptoms. Scores range from 0-36 with higher scores reflecting greater symptom severity.
Mean change score in Generalized Anxiety Disorder Scale (GAD-7) | Change at 2-month follow-up from baseline
  The 7-item GAD-7 measures severity of anxiety symptoms. Scores range from 0-28 with higher scores reflecting greater symptom severity.
Mean change score in McGill Pain Questionnaire | Change at 2-month follow-up from baseline
  The McGill Pain Questionnaire assesses pain intensity and type. Scores range from 0-100 with higher scores reflecting greater pain severity.
Mean change in Short Form Veteran Health Survey (VR-12) | Change at 2-month follow-up from baseline
  The VR-12 is a short-form measures self-reported health and functioning. Higher scaled scores indicate greater functional impairment.

OTHER OUTCOMES:
Mean change score in Chronic Pain Acceptance Questionnaire (CPAQ-Revised) | Change at 2-month follow-up from baseline
  The 20-item CPAQ-revised is designed to measure acceptance of pain, which is thought to reduce unsuccessful attempts to avoid or control pain and thus focus on engaging in valued activities and pursuing meaningful goals. Scores range from 0-120 with higher scores reflecting greater pain acceptance.
Mean change score in Chronic Pain Values Inventory (CPVI) | Change at 2-month follow-up from baseline
  The 12-item CPVI measures which values are important to an individual and the degree of success they are having in following their values. Two average scores are created (mean success and mean discrepancy ratings) that range from 0-5. Higher mean scores reflect greater success or greater discrepancy between importance of value and success in achieving it.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States